CLINICAL TRIAL: NCT01785160
Title: Investigation of Faldaprevir Effect on Steady State Pharmacokinetics of Raltegravir in Healthy Male and Female Volunteers (an Open-label Trial With Two Periods in a Fixed Sequence)
Brief Title: Investigation of Faldaprevir Effect on Pharmacokinetics of Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1220.65; 2012-004872-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-12-13; First posted 2013-02-07 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — Raltegravir Potassium; faldaprevir

ARMS (2):
- Raltegravir (Active Comparator): coated tablets, oral administration with 240 ml water
  Interventions: Drug: Raltegravir
- Raltegravir + Faldaprevir (Experimental): coated tablets and soft gelatine capsule, oral administration with 240 ml water
  Interventions: Drug: Raltegravir; Drug: Faldaprevir

INTERVENTIONS:
Drug: Raltegravir — low dose oral administration
  Arms: Raltegravir
Drug: Raltegravir — low dose oral administration
  Arms: Raltegravir + Faldaprevir
Drug: Faldaprevir — medium dose oral administration
  Arms: Raltegravir + Faldaprevir

SUMMARY:
The primary objective of this trial is to investigate effect of faldaprevir on steady state pharmacokinetics of raltegravir.

The assessment of safety and tolerability will be an additional objective of this trial.

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.65.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Total number of patients randomised and treated in the study.This was a open label trial with two periods in a fixed sequence. All subjects were to receive the following 2 treatments, A]Raltegravir B]Raltegravir+Faldaprevir. The two treatments were separated by washout period of at least 7 days.
Period: Treatment Period 1: Raltegravir
Arm/Group | Overall Study
Started | 25
Completed | 24
Not Completed | 1
Not completed — Not treated | 1
Period: Washout Period of at Least 7 Days
Arm/Group | Overall Study
Started | 24
Completed | 23
Not Completed | 1
Not completed — Consent withdrawn | 1
Period: Treatment Period 2: Raltegravir + Faldap
Arm/Group | Overall Study
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The total number of participants N analysed for baseline characteristics is not same as the number of participants enrolled as one subject was not treated after being enrolled
Groups:
- Overall Study: Total number of patients randomised and treated in the study.This was a open label trial with two periods in a fixed sequence. All subjects were to receive the following 2 treatments, A]Raltegravir B]Raltegravir+Faldaprevir The two treatments were separated by washout period of at least 7 days.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: AUC( Tau,ss)
Description: AUC tau,ss (area under the concentration-time curve of the Raltegravir in plasma at steady state over the uniform dosing interval tau) Point estimates for the intrasubject ratio of the geometric means (for treatments Test and Reference) of AUC tau,ss and their 2-sided 90% confidence intervals (CI) were calculated.
  The statistical model was an analysis of variance (ANOVA) on log-transformed parameters including effects for 'subject' and 'treatment'.
  RAL: Raltegravir , FDV: Faldaprevir
Time Frame: 0.5 hours (h) before drug administration and 48 hours (h),60,72,72.5,73,73.5,74,75,76,77,78,80,82 and 84(hours) after administration of RAL alone; 96 h,108,120,120.5,121,121.5,122,123,124, 125,126,128,130 and 132 hours after RAL and FDV administration
Population: Pharmacokinetic(PK) set:Subjects who received atleast 1 dose of study medication and who provided at least 1 observation for at least 1 PK endpoint without any important protocol violations relevant to the evaluation of relative bioavailability and did not experience emesis at or before 2 times median tmax on the pk study days of both trial periods
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Raltegravir: Raltegravir coated tablets
  Oral with 240 mL of water Days 1 to 3: 400 mg raltegravir twice daily Day 4: 400 mg raltegravir once daily
- Raltegravir + Faldaprevir: Raltegravir coated tablets and Faldaprevir soft gelatin capsules
  Oral with 240 mL of water Day 1: 400 mg raltegravir twice daily and 240 mg faldaprevir twice daily (loading dose) Days 2 to 5: 400 mg raltegravir twice daily and 240 mg faldaprevir once daily Day 6: 400 mg raltegravir once daily and 240 mg faldaprevir once daily
Arm/Group | Raltegravir | Raltegravir + Faldaprevir
Number analyzed (Participants) | 24 | 23
ng*h/mL | 4070 (92.9) | 11100 (78.7)
Statistical Analysis 1: Comparison: Raltegravir vs Raltegravir + Faldaprevir; Ratio Raltegravir plus Faldaprevir and Raltegravir for the category Raltegravir; Test type: Non-Inferiority or Equivalence — Relative bioavailability (No formal testing was performed); p = 0.9999, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted Geometric Mean ratio = 272.06, 95% CI [199.69 to 370.66], Standard Deviation 67.9 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cmax ,ss
Description: C max,ss (maximum measured concentration of the Raltegravir in plasma at steady state) Point estimates for the intrasubject ratio of the geometric means (for treatments Test and Reference) of Cmax,ss and their 2-sided 90% confidence intervals (CI) were calculated.
  The statistical model was an analysis of variance (ANOVA) on log-transformed parameters including effects for 'subject' and 'treatment'.
  RAL: Raltegravir , FDV: Faldaprevir
Time Frame: 0.5 hours (h) before drug administration and 48 hours (h),60,72,72.5,73,73.5,74,75,76,77,78,80,82 and 84(hours) after administration of RAL alone; 96 h,108,120,120.5,121,121.5,122,123,124, 125,126,128,130 and 132hours after RAL and FDV administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Raltegravir | Raltegravir + Faldaprevir
Number analyzed (Participants) | 24 | 23
ng/mL | 1300 (115) | 3220 (108)
Statistical Analysis 1: Comparison: Raltegravir vs Raltegravir + Faldaprevir; Ratio Raltegravir plus Faldaprevir and Raltegravir for the category Raltegravir; Test type: Non-Inferiority or Equivalence — Relative bioavailability(No formal testing was performed); p = 0.9973, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted Geometric Mean ratio = 245.72, 95% CI [168.460 to 358.404], Standard Deviation 87.1 — The standard deviation is actually the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: Up to 23 days (+1day)
Arm/Group | Raltegravir | Raltegravir + Faldaprevir
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 6/24 | 13/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir (N=24) | Raltegravir + Faldaprevir (N=23)
Headache (Nervous system disorders) | 3 | 5
Dizziness (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.